CLINICAL TRIAL: NCT06300515
Title: Physical Exercise and Health Counseling in Patients With Pediatric Cancer Patients Undergoing Hematopoietic Stem Cell Transplantation: From Research to Clinical Reality.
Brief Title: Exercise and Health Counseling in Pediatric Hematopoietic Stem Cell Transplantation
Acronym: HENKO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alejandro Lucia (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor-Investigator, Alejandro Lucia, Professor, Universidad Europea de Madrid
Organization: Universidad Europea de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PI23/00396
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hematopoietic System--Cancer
Keywords: exercise; pediatric cancer; health counseling
MeSH Terms: conditions — Motor Activity; Neoplasms | interventions — Control Groups; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The staff in charge of outcome assessment will be blinded to the group assigned to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): During the intervention phase (hospitalization for hematopoietic stem cell transplantation (HSCT) and subsequent 8-week outpatient phase following discharge), the control group will participate in a Health Counseling Program (1 time/week) on aspects related to a healthy lifestyle such as reducing sedentary lifestyle, acquiring healthy nutritional habits, the importance sleep, screen use, and how to address barriers related to clinical status. We will adapt the program to the needs and timing of the patient's treatment, providing the content in one session/week orally (e.g. using presentations) and in writing (e.g. through brochures).
  Interventions: Behavioral: Control Group (Active Comparator)
- Exercise (Experimental): During the intervention phase (hospitalization for hematopoietic stem cell transplantation (HSCT) and subsequent 8-week outpatient phase following discharge), the intervention group will participate in exactly the same Health Counseling Program as the Control group. Additionally, this group will perform an exercise program combining aerobic and muscle strength exercises
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Control Group (Active Comparator) — During the intervention phase (hospitalization for HSCT and subsequent 8-week outpatient phase following discharge), the control group will participate in a Health Counseling Program (1 time/week) on aspects related to a healthy lifestyle such as reducing sedentary lifestyle, acquiring healthy nutritional habits, the importance sleep, screen use, and how to address barriers related to clinical status. We will adapt the program to the needs and timing of the patient's treatment, providing the content in one session/week orally (e.g. using presentations) and in writing (e.g. through brochures).
  Other Names: Health Counseling only
  Arms: Control
Behavioral: Intervention Group — Same as Control Group + exercise program as described below:
  Same as Control Group + exercise program as described below:
  Hospital ward (during HSCT); and Hospital Gym or online (patients' home) during the outpatient phase. Frequency: 3-5 days/week. Session duration: 30 to 55-60 minutes Aerobic training (5-25 minutes): bicycling, crank-ergometry, circuit-style exercises, and games. Muscle strength training (10-20 minutes): large muscle group exercises (upper/lower limb + trunk exercises) performed as a circuit using body weight or against resistance (against gravity and with body weight, elastic bands, dumbbells, weighted vests, machines), with a wide range of joint mobility and at submaximal/maximum voluntary speed. Inspiratory muscle training will also be performed (5 min daily, using a specific device that creates resistance against inspiration).
  Other Names: Health Counseling + Exercise
  Arms: Exercise

SUMMARY:
Thanks to medical advances, survival rates >5 years in children/adolescents undergoing hematopoietic stem cell transplant (HSCT) exceed 70%. However, these patients are at high risk of suffering sequelae associated with the underlying disease and/or the HSCT itself, which negatively affects their physical capacity. These patients also tend to spend too much time inactive, which further accelerates functional decline in addition to producing fatigue and impairing quality of life. Therefore, new strategies are needed to minimize the morbidity associated with HSCT. In this effect, although physical exercise represents an interesting adjuvant treatment option for HSCT, scientific evidence in this area is still scarce. Implementation of physical exercise intervention in pediatric HSCT units is challenging due to the lack of research on the effectiveness, affordability and accessibility of this type of intervention. Therefore, establishing the effectiveness of physical exercise under controlled conditions is an important step. The investigators therefore aim to assess the impact of a physical exercise and health counseling program, compared to health counseling only (control group), in pediatric patients with cancer undergoing HSCT on physical-functional, behavioral, psycho-cognitive and clinical outcomes, and blood biomarkers. The investigators will also determine to what extent the benefits of this intervention are maintained over time. Additionally, the investigators will determine the feasibility of implementing the proposed intervention in a real clinical situation in 3 different pediatric HSCT units.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT), which is used to treat high-risk malignancies, as well as some other conditions or even autoimmune processes, consists of several phases: mobilization and subsequent collection of hematopoietic stem cells from the patient (autologous HSCT) or from a donor (allogeneic HSCT); pre-HSCT conditioning; infusion of patient/donor cells; establishment of a new immune and hematopoietic system in the recipient; and prophylaxis/treatment of possible adverse effects. Since the first successful allogeneic transplant was performed in 1968, thanks to the advances experienced in conditioning regimens, as well as in donor-recipient histocompatibility testing, in patient care and in the management of graft versus host disease (GvHD), together with the increase in the number of donors, the expectations of children and adolescents who receive HSCT have improved, achieving long-term survival rates (>5 years) >70%. Yet survivors are at high risk of suffering side effects and toxicities derived from the HSCT itself and/or the underlying disease, with subsequent functional decline. In addition, they show a higher risk of rehospitalization than pediatric cancer survivors who did not receive HSCT and tend to develop chronic pathologies (especially cardiometabolic conditions and frailty) at earlier stages of adulthood than the general population.

The investigators therefore aim to assess the impact of a physical exercise and health counseling program, compared to health counseling only (control group), in pediatric patients with cancer undergoing HSCT on the following outcomes assessed at 3 time points [start of hospitalization for HSCT (i.e., baseline), and 8 weeks and 3 months after hospital discharge, respectively]: cardiorespiratory fitness (primary outcome) and ventilatory threshold, muscle strength, left ventricle ejection fraction, fractional shortening and global longitudinal strain, total cardiac mass, functional mobility, adiposity (waist to hip ratio), body mass index, dual-energy X-ray absorptiometry (DXA)-determined body composition (lean and fat mass, bone mineral density), accelerometry-determined physical activity levels, ankle dorsiflexion range of motion, health-related quality of life, cancer-related fatigue, and immune subpopulations. We will also determine clinical outcomes during hospitalization (survival, treatment tolerability, toxicities) as well as molecular biomarkers in blood.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 and 21 years.
* Undergoing hematopoietic stem cell transplantation (HSCT) for cancer diagnosis in complete remission or without remission, in 3 recruiting Hospitals in Madrid
* Undergoing treatment and follow-up in the same hospital.
* Speaking Spanish.
* Providing signed informed consent.

Exclusion Criteria:

* Not being able to participate in the trial according to protocol.
* Comorbidity or acute condition not associated with the diagnosis and that contraindicates the practice of physical exercise, such as severe deficiencies in the locomotor, neurological, cardiovascular and pulmonary systems.
* Serious or chronic medical or psychiatric condition that may increase the risk associated with participation in the trial or that may interfere with the interpretation of the results and, in the opinion of the investigator in discussion with the team, makes having such condition inappropriate for entry to this study; inability to understand the study requirements.
* Not being able to attend hospital visits to perform assessment tests, nor participate in the physical exercise and health counseling program as stipulated in the protocol.

Inability to understand the requirements of the study.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in objectively-assessed cardiorespiratory fitness (CRF) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  CRF assessed as peak oxygen uptake, as determined during a ramp bicycle ergometer test until volitional exhaustion (unit = mL of oxygen/kg body mass/minute),
Change in estimated cardiorespiratory fitness (CRF) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  CRF estimated with 6-minute walking distance (maximum distance achieved) (unit = meters)

SECONDARY OUTCOMES:
Change in isometric leg muscle strength from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Dynamometer-determined maximal isometric strength of knee flexor muscles (unit = Newtons)
Change in dynamic lower-limb muscle strength from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  One-repetition maximum (1RM) during leg press exercise, as estimated from 5RM leg press (unit = kg)
Change in upper-limb muscle strength from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Maximal handgrip strength, mean of 3 attempts with both arms (unit = kg)
Change in respiratory muscle strength from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Maximal inspiratory pressure (unit = mm H20)
Change in the 'ventilatory threshold' (VT) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Workload eliciting the ventilatory threshold, as determined during the ramp test (unit = watts)
Change in left ventricle (LV) ejection fraction from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Echocardiography-determined LV ejection fraction (unit = percent)
Change in left ventricle (LV) fractional shortening from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Echocardiography-determined LV fractional shortening (unit = percent)
Change in left ventricle (LV) global longitudinal strain (GLS) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Echocardiography-determined GLS of the LV (unit = percent)
Change in total cardiac mass from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Echocardiography-determined total cardiac mass (unit = grams divided by body surface area (im meters squared)
Change in functional mobility (stairs test) from baseline to follow-uo | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Stairs test (time to walk up and down a 12-step stair) (unit = seconds)
Change in functional mobility (chair rising) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Sit-stand test (time to stand from a chair 5 times) (unit = seconds)
Change in functional mobility (Quick Function test) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  We will use the Quick Motor Function test, which takes approximately 10 to 15 minutes. An evaluator observes the performance of a patient and scores the 16 items separately on a 5-point ordinal scale (ranging from 0 to 4). If items can be performed on both left and right extremities, the right side is taken. A total score is obtained by adding the scores of all items. The total score ranges between 0 and 64 points (units = points, from 0 to 64)
Change in body mass index (BMI) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  BMI is measured as weight (kg) divided by height squared (m2)
Change in adiposity index from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Waist-to-hip ratio (no units)
Change in dual-energy X-ray absorptiometry (DXA) measures of total lean mass from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  DXA-determined total lean mass (grams)
Change in dual-energy X-ray absorptiometry (DXA) measures of total fat mass from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  DXA-determined total fat mass (grams)
Change in dual-energy X-ray absorptiometry (DXA) measures of bone health from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  DXA-determined bone mineral density (unit = grams/m2)
Change in physical activity (PA) from baseline to end of treatment | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  PA levels (moderate/vigorous PA) determined using triaxial accelerometry (unit = minutes/week)
Change in ankle-dorsiflexion from baseline to end of treatment | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Goniometer-determined active and passive ankle range of motion in dorsiflexion (unit = degrees)
Change in psychological status (health-related quality of life) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Health-related QoL (HRQoL) (Paediatric Quality of Life Inventory [abbreviated as PedsQL 4.0] Cancer Module [3.0], designed to measure paediatric/adolescent cancer specific HRQoL) (unit = 0 to 100 scale, with higher scores indicating better HRQoL)
Change in psychological status (fatigue) from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Cancer-related fatigue (Paediatric Quality of Life (PedsQL 3.0) Multidimensional Fatigue Scale) (0 to 100 score, higher scores meaning higher fatigue)
Change in lymphocyte subpopulations from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Flow-cytometry determined lymphocyte subpopulations (unit = %)
Change in immune phenotype from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Flow-cytometry determined natural killer (NK) cell subsets (unit = %)
Change in survival from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Survival (number of days from diagnosis to the end of the study or death)
Change in treatment tolerability from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Treatment interruption/delay (number of days)
Change in treatment toxicities from baseline to follow-up | Assessed at three time points: (1) start of hospitalization for HSCT (i.e., baseline); (2) 8 weeks after hospital discharge; and (3) 3 months after hospital discharge (i.e., follow-up)
  Common Toxicity Criteria for Adverse Events [CTCAE, global score, 1 (low toxicity) to 5 (highest])
Change in the 'acute' molecular response to a single exercise session from baseline to 8 weeks after hospital discharge | Assessed at two time points: (1) start of hospitalization for HSCT (i.e., baseline); and (2) 8 weeks after hospital discharge.
  Panel of cytokines/chemokines and peptides (oncostatin-M, osteonectin, FGF21, irisin, follistatin-1, musclin, VEGF-A, fractalkine, interleukin (IL)-8, IL-6 and IL-15 in serum using Luminex® (all assessed in the same units, micrograms/dL) before and after a single exercise training session
Change in the 'chronic' (resting conditions) transcriptome from baseline to 8 weeks after hospital discharge | Assessed at two time points: (1) start of hospitalization for HSCT (i.e., baseline); and (2) 8 weeks after hospital discharge.
  RNA sequencing (RNAseq) profile in peripheral blood mononuclear cells under resting conditions at baseline and 8 weeks after hospital discharge
Change in the 'acute' transcriptome response to a single exercise session from baseline to 8 weeks after hospital discharge | Assessed at two time points: (1) start of hospitalization for HSCT (i.e., baseline); and (2) 8 weeks after hospital discharge.
  RNA sequencing (RNAseq) profile in peripheral blood mononuclear cells before and after a single exercise training session
Change in the 'acute' transcriptome response from baseline to 8 weeks after hospital discharge | Assessed at two time points: (1) start of hospitalization for HSCT (i.e., baseline); and (2) 8 weeks after hospital discharge.
  RNA sequencing (RNAseq) profile in peripheral blood mononuclear cells before and after and exercise training session

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital 12 de Octubre, Madrid, Spain